CLINICAL TRIAL: NCT05050929
Title: Randomized Phase II Non-Inferiority Study of 5-Day Versus 1-Day RAPid SimPLE (RAPPLE) Targeted Radiation Treatment for Brain Metastases
Brief Title: RAPid SimPLE Targeted Radiation Treatment for Brain Metastases
Acronym: RAPPLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-01343
Record Dates: First submitted 2021-08-04; First posted 2021-09-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Brain Metastases, Adult
Keywords: radiotherapy; randomized clinical trial; phase II; non-inferiority; overall survival
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Equal arms (1:1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 20 Gy in 5 Fractions Volumetric Modulated Arc Therapy to Brain Metastases (Active Comparator): Five treatments of 4 Gy will be delivered using volumetric modulated arc therapy on a conventional linear accelerator in a conventional head shell without the use of stereotactic radiosurgery technique.
  Interventions: Radiation: Targeting All Brain Metastases
- 8 Gy in 1 Fraction Volumetric Modulated Arc Therapy to Brain Metastases (Experimental): A single treatment of 8 Gy will be delivered using volumetric modulated arc therapy on a conventional linear accelerator in a conventional head shell without the use of stereotactic radiosurgery technique.
  Interventions: Radiation: Targeting All Brain Metastases

INTERVENTIONS:
Radiation: Targeting All Brain Metastases — Volumetric Modulated Arc Therapy

SUMMARY:
The aim of the study is to show that rapid, simple targeted radiotherapy to brain metastases with 8 Gy / 1 is non-inferior to 20 Gy / 5 in terms of overall survival for patients with poor prognosis.

DETAILED DESCRIPTION:
Hypothesis For selected patients with limited life expectancy, a single targeted fraction of 8 Gy / 1 to brain metastases will provide equivalent survival as targeted radiotherapy with 20 Gy / 5 to brain metastases.

Justification The QUARTZ study randomized patients with brain metastases and poor prognosis between 20 Gy / 5 whole brain radiotherapy (WBRT) and best supportive care. The median survival in both arms of the study was 9 weeks. The quality of life in both arm was also the same. It is known that WBRT significantly diminishes quality of life. The investigators interpretation of the QUARTZ trial is that the unchecked growth of brain metastases in the best supportive care arm diminishes quality of life as much as WBRT. To control brain metastases without giving WBRT, targeted treatment with 20 Gy / 5 to the metastases alone is standard care at BC Cancer. Numerous randomized trials have compared the efficacy of 20-30 Gy / 5-10 fractions and 8 Gy / 1 for palliative treatment of pain from bone metastases. In addition, there is a randomized trial showing that 20 Gy / 5 and 8 Gy /1 are equally effective for the treatment of symptoms from spinal cord compression. This study will test the use of this shorter, one-visit treatment schedule against the standard 5-visit treatment schedule for patients with brain metastases.

Research Design Randomized Phase II Non-Inferiority Study. The estimated median survival for this cohort, based upon a prior cohort study from 2012-2016 at BC Cancer is 3 months (13 weeks). The investigators would regard a study median survival of less than the 9-week median survival observed in the QUARTZ trial as unacceptable. Hence, the hazard ratio for the experimental arm and the control arm is: 13 weeks / 9 weeks = 1.44. With one-sided Type I error set at alpha = 0.2 and power = 0.8, the investigators calculated a theoretical sample size of 86 patients. Based on prior experience with clinical trials for patients with brain metastases, a 15% risk of drop-out and loss to follow up is expected. Hence the final sample size will be 100 patients. Stratification by the diagnosis-specific graded prognostic assessment (DS-GPA) ranges of 0.0 - 1.0 and 1.5 - 2.0 and lung cancer versus other histologies will help to ensure baseline characteristics that predict for equal survival are equally distributed in both arms of the study.

Statistical Analysis The primary endpoint is overall survival. The study will be considered to be a positive phase II non-inferiority study if the median survival in the experimental arm is within 4 weeks of the median survival in the standard arm.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for participation in this study:

* Age ≥ 18
* Pathological diagnosis of a non-hematopoietic malignancy
* Brain metastases of any size
* Any number of untreated or progressing, previously treated brain metastases that can all be contoured and targeted
* Presence of extracranial disease
* Diagnosis-Specific Graded Prognostic Assessment ≤ 2.0. (https://brainmetgpa.com/) or Graded Prognostic Assessment ≤ 2.0 (Appendix I)
* Able to complete the EuroQOL (EQ-5D-5L) questionnaire
* Willing and able to have regular imaging follow up
* Feasible to start protocol treatment within 14 days of participant enrolment
* Karnofsky Performance Score (KPS) ≥ 50

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

* Inability to have a brain MRI
* WBRT less than 3 months prior to randomization
* Disseminated leptomeningeal carcinomatosis (limited pachymeningeal disease is permitted)
* Multiple sclerosis
* Neurologically declining despite corticosteroids
* Appropriate for surgery or stereotactic radiosurgery
* Germ cell and primary brain tumours
* Systemic lupus erythematosis, scleroderma, or other connective tissue disorders not in remission
* Any other serious intercurrent illness or medical condition judged by the local investigator to compromise the participant's safety, preclude safe administration of the planned protocol treatment, or prevent the participant from being managed according to the protocol guidelines
* Pregnancy
* Potentially fertile men or women of childbearing potential who are unwilling to employ highly effective contraception

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival Time | 1 year
  The median time from randomization to death

SECONDARY OUTCOMES:
Median Time to Decline in Karnofsky Performance Status | 1 year
  The time from randomization to a 20-point decline in Karnofsky Performance Status
Control of treated brain metastases | 1 year
  Cumulative incidence of local recurrence of treated metastases
Corticosteroid use | 6 weeks
  Proportion of patients taking corticosteroids
Control of brain disease | 1 year
  Cumulative incidence of (local recurrence of treated metastases OR new metastases)
Retreatments for brain metastases | 1 year
  Proportion of patients with retreatment for brain metastases after radiotherapy
Adverse Events | 1 year
  Cumulative incidence of adverse events, graded using CTCAE Version 5.0
Health-Related Quality of Life | 1 year
  Median time to a minimum clinically important decline in Health-Related Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Alan Nichol, MD, Principal Investigator — BC Cancer Vancouver
Locations (6):
- Canada (6):
  - BC Cancer - Abbotsford, Abbotsford, British Columbia
  - BC Cancer - Kelowna, Kelowna, British Columbia
  - BC Cancer - Prince George, Prince George, British Columbia
  - BC Cancer - Surrey, Surrey, British Columbia
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia

REFERENCES:
- [Background] Mulvenna P, Nankivell M, Barton R, Faivre-Finn C, Wilson P, McColl E, Moore B, Brisbane I, Ardron D, Holt T, Morgan S, Lee C, Waite K, Bayman N, Pugh C, Sydes B, Stephens R, Parmar MK, Langley RE. Dexamethasone and supportive care with or without whole brain radiotherapy in treating patients with non-small cell lung cancer with brain metastases unsuitable for resection or stereotactic radiotherapy (QUARTZ): results from a phase 3, non-inferiority, randomised trial. Lancet. 2016 Oct 22;388(10055):2004-2014. doi: 10.1016/S0140-6736(16)30825-X. Epub 2016 Sep 4. PMID 27604504